CLINICAL TRIAL: NCT04359186
Title: Analytic Treatment Interruption in HIV Infection
Brief Title: SCOPE Analytic Treatment Interruption Protocol
Acronym: SCOPE-ATI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Chan Zuckerberg Biohub (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-30442
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS
Keywords: HIV; HIV/AIDS; Antiretroviral therapy; HIV reservoir; Biomarkers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Interruption Arm (Experimental)
  Interventions: Other: Treatment Interruption Arm

INTERVENTIONS:
Other: Treatment Interruption Arm — Individuals with HIV on suppressive ART will interrupt their ART.

SUMMARY:
The goal of this study is to understand the interaction between HIV and the host at the earliest stages when HIV medications are paused. Volunteers with HIV will interrupt antiretroviral therapy (ART) and then have intensive studies preformed two to three times per week. Most will resume therapy within three weeks, even if the virus does not rebound during this time.

DETAILED DESCRIPTION:
In this study, people living with HIV will undergo intensive sampling prior to and following an interruption of their antiretroviral therapy (ART). Individuals will be asked to resume ART once the virus is detectable, or after approximately three weeks if the virus remains undetectable.

Individuals who were able to control their virus before ART ("controllers") will be able to participate in an extended treatment interruption and have less restrictive ART restart criteria.

The overall goal of the study is to characterize the interaction between the host and the virus at the earliest stages of virus replication and to identify predictors of rebound before virus becomes detectable.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age >= 18
* Documented HIV infection
* Antiretroviral therapy for at least 12 months
* Screening plasma HIV RNA levels below level of detection (< 40-75 copies/mL), and all available determinations in past 12 months also below level of detection (blips allowed)
* Screening CD4+ T-cell count >350 cells/uL
* If of childbearing potential, willing to use two methods of contraception
* Willing to receive counseling regarding HIV transmission risk mitigation

Exclusion Criteria:

* Pregnant or plans to become pregnant during the course of the study
* Active hepatitis B, defined as (1) positive sAg or (2) positive cAb with negative sAb and positive HBV DNA
* Active hepatitis C, defined as positive Hep C Ab with positive HCV RNA
* Use of a non-nucleoside reverse transcriptase inhibitor and unable to switch regimen
* Significant cardiovascular or cerebrovascular disease
* Recent or prior (within past 5 years) malignancy
* Severe kidney disease (CrCl < 50 mL/min via Cockroft-Gault method)
* Severe hepatic impairment (Child-Pugh Class C) or unstable liver disease
* Concurrent treatment with immunomodulatory drugs
* Unable or unwilling to use barrier protection or pre-exposure prophylaxis (PrEP) to prevent HIV transmission with sexual partners not known to be HIV-infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Acute retroviral syndrome | Week 0 through Month 6
  The proportion of participants developing acute retroviral syndrome
Failure to re-suppress | Week 0 through Month 12
  The proportion of participants who fail to re-suppress to plasma HIV RNA levels <50 copies/mL after re-initiating ART
CD4+ T cell decline | Week 0 through Month 6
  The proportion of participants with confirmed decreases in CD4+ T cell count below 350 cells/uL
Time to rebound | Week 0 through Month 6
  The time between the treatment interruption and plasma HIV RNA >200 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No